CLINICAL TRIAL: NCT01193348
Title: An Open-Label, Multi-Center Clinical Trial of Eculizumab in Pediatric Patients With Atypical Hemolytic-Uremic Syndrome
Acronym: aHUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C10-003
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Results first posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Atypical Hemolytic-Uremic Syndrome
Keywords: Atypical Hemolytic-Uremic Syndrome
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eculizumab (Experimental)
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Fixed dosing is based on body weight cohorts. Adjustment of dose to accommodate patient growth is possible.

SUMMARY:
The primary purpose is to assess the efficacy and safety of eculizumab in pediatric patients with aHUS to control TMA as characterized by thrombocytopenia, hemolysis and renal impairment.

ELIGIBILITY:
Inclusion:

1. Patient's parent/legal guardian must have been willing and able to give written informed consent and the patient must have been willing to give written informed assent (if applicable as determined by the central IRB/IEC).
2. Pediatric patients with aHUS: Patients could have been newly diagnosed, or with previously diagnosed disease, or post-kidney transplant with the disease.
3. Patients one month to 18 years and body weight ≥ 5kg.
4. Platelet count at screening and baseline visit must have been below lower limit of normal (<LLN). If screening visit and baseline visit are combined into one day, an additional platelet count value obtained at least 24 hours before screening/baseline sample must also be <LLN.
5. Exhibited signs or symptoms of hemolysis at start of current aHUS event (i.e., lactate dehydrogenase (LDH) ≥1.5 x Upper Limit of Normal [ULN] and hemoglobin ≤LLN), fragmented RBC with a negative Coombs test.
6. Serum Creatinine level ≥97 percentile for age at screening (patients requiring dialysis for acute renal failure are also eligible).
7. Patients with aHUS due to complement regulatory protein genetic abnormality or anti-complement factor antibody or those in whom known etiologies of hemolytic uremic syndrome (HUS) have been ruled out as confirmed in the Exclusion Criteria.
8. Patients must have been vaccinated against N. meningitidis, pneumococcus and haemophilus (per the vaccine label) at least 14 days prior to study drug initiation or otherwise be protected by prophylactic antibiotics. Patients under age two years were to receive antibiotic prophylaxis throughout the treatment period.
9. Female patients of childbearing potential (female patients who have achieved menarche) must have been practicing an effective, reliable and medically approved contraceptive regimen during the entire duration of the study, including the follow-up period. At the time of the last follow-up visit, patients must have agreed to continue to use adequate contraception methods for up to five months following discontinuation of eculizumab treatment.
10. Able and willing to comply with study procedures

Exclusion:

Any of the following was regarded as a criterion for exclusion from the study:

1. Known familial ADAMTS-13 deficiency (ADAMTS-13 <5%).
2. Shiga toxin E.coli-related hemolytic uremic syndrome (STEC-HUS [known Shiga toxin + E.coli]).
3. History of malignancy within five years of screening.
4. Known human immunodeficiency virus (HIV) infection.
5. Identified drug exposure-related HUS.
6. Infection-related HUS.
7. HUS related to bone marrow transplant (BMT).
8. HUS related to vitamin B12 deficiency.
9. Known Systemic Lupus Erythematosus (SLE) or antiphospholipid antibody positivity or syndrome.
10. Plasma Therapy for >5 weeks prior to enrollment.
11. Chronic dialysis (defined as dialysis on a regular basis as renal replacement therapy for end-stage renal disease [ESRD]).
12. Patients with a confirmed diagnosis of sepsis defined as positive blood cultures within seven days of the screening visit and not treated with antibiotics to which the organism is sensitive.
13. Presence or suspicion of active and untreated systemic bacterial infection that, in the opinion of the Investigator confounds an accurate diagnosis of aHUS or impedes the ability to manage the aHUS disease.
14. Pregnancy or lactation.
15. History of meningococcal/pneumococcal/gonococcal disease.
16. Any medical or psychological condition that, in the opinion of the investigator, could increase the patient's risk by participating in the study or confound the outcome of the study.
17. Patients receiving chronic intravenous immunoglobulin (IVIg) within eight weeks unless for unrelated medical condition (e.g., Hypogammaglobinemia), or chronic Rituximab therapy within 12 weeks of the screening visit.
18. Patients receiving other immunosuppressive therapies such as steroids, mTOR inhibitors, calcineurin inhibitors (e.g., cyclosporine or tacrolimus are excluded unless: [1] part of an established post-transplant anti-rejection regime, or [2] patient has confirmed anti-Complement Factor antibodies antibody requiring immunosuppressive therapy or [3] steroids are being used for a condition other than aHUS (example asthma).
19. Participation in any other investigational drug trial or device trial, or procedures beginning four weeks prior to screening and throughout the entire trial
20. Prior use of eculizumab, hypersensitivity to eculizumab, to murine proteins or to one of the excipients.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2010-09; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (4):
  - Atlanta, Georgia
  - Hackensack, New Jersey
  - Corpus Christi, Texas
  - Spokane, Washington
- North Adelaide, South Australia, Australia
- Ghent, Belgium
- Toronto, Ontario, Canada
- France (4):
  - Lille
  - Marseille
  - Paris
  - Rouen
- Hanover, Germany
- Italy (2):
  - Milan
  - Palermo
- Nijmegen, Netherlands
- United Kingdom (2):
  - London
  - Nottingham

REFERENCES:
- [Derived] Pugh D, O'Sullivan ED, Duthie FA, Masson P, Kavanagh D. Interventions for atypical haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2021 Mar 23;3(3):CD012862. doi: 10.1002/14651858.CD012862.pub2. PMID 33783815
- [Derived] Tschumi S, Gugger M, Bucher BS, Riedl M, Simonetti GD. Eculizumab in atypical hemolytic uremic syndrome: long-term clinical course and histological findings. Pediatr Nephrol. 2011 Nov;26(11):2085-8. doi: 10.1007/s00467-011-1989-4. Epub 2011 Aug 30. PMID 21877169

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 27 patients diagnosed with aHUS signed the informed consent and of these, 22 patients were treated. Five patients were excluded from the study due to failed screening procedure and did not receive eculizumab.
Pre-assignment Details: At screening, patients had to have a platelet count < lower limit of normal range (<LLN) and serum creatinine level > 97 percentile for age; and had to exhibit signs or symptoms of hemolysis at the start of the current aHUS event with fragmented RBC and a negative Coombs test.
Period: Screening Period
Arm/Group | Eculizumab
Started | 27
Completed | 22
Not Completed | 5
Not completed — Screen Failure | 5
Period: Treatment Period (26 Weeks)
Arm/Group | Eculizumab
Started | 22
Completed | 19
Not Completed | 3
Not completed — Positive Shiga-Toxin Result vial Local | 1
Not completed — Serious Adverse Event | 1
Not completed — Patient Requested to Withdraw | 1
Period: Extension Treatment Period
Arm/Group | Eculizumab
Started | 17
Completed | 16
Not Completed | 1
Not completed — Physician Decision | 1
Period: Post Treatment Period (Patients Who Disc
Arm/Group | Eculizumab
Started | 10
Completed | 8
Not Completed | 2
Not completed — Patient did not return for visit | 2

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population was defined as all patients who received any amount of eculizumab, and were considered evaluable for safety and efficacy analyses. For both the efficacy and safety analyses, all 22 patients who were treated with study drug were included in the ITT population.
Arm/Group | Eculizumab
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.6 (6.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Complete TMA Response
Description: Proportion of Patients with Complete TMA response was determined and defined by normalization of hematological parameters (platelet count and LDH) and ≥ 25% improvement in serum creatinine from baseline which was sustained for at least two consecutive measurements obtained at least four weeks apart).
Time Frame: Through 26 weeks
Population: The tabulations of the proportions of patients with Complete TMA Response through 26 weeks were performed for the ITT population. Exact binomial two-sided 95% CI using the Clopper-Pearson method for the responder rate was presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 22
Percentage of Participants | 63.6 [40.7 to 82.8]
Statistical Analysis 1: Comparison: Eculizumab; Test type: Superiority or Other; Percent of Complete TMA Response = 63.6, 95% CI 2-sided [40.7 to 82.8]

2. Secondary Outcome: Proportion of Patients With Complete Hematologic Response
Description: Proportion of Patients with Complete Hematologic response through 26 weeks of treatment was determined and defined by normalization of platelet count and LDH sustained for at least two consecutive measurements obtained at least four weeks apart.
Time Frame: Through 26 weeks
Population: The tabulations of the proportions of patients with Complete Hematologic Response through 26 weeks were performed for the ITT population. The number of patients with response and responder rate, along with an exact two-sided 95% CI were summarized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 22
Percentage of Participants | 81.8 [59.7 to 94.8]
Statistical Analysis 1: Comparison: Eculizumab; Test type: Superiority or Other; Percent of Complete Hematologic Response = 81.8, 95% CI 2-sided [59.7 to 94.8]

3. Secondary Outcome: Proportion of Patients With Platelet Count Normalization
Description: Proportion of Patients with Platelet Count Normalization through 26 weeks of treatment was determined and defined as the platelet count observed to be ≥ 150 x 109/L on at least two consecutive measurements which span a period of at least four weeks.
Time Frame: Through 26 weeks
Population: The tabulations of the proportions of patients with Platelet Count Normalization through 26 weeks were performed for the ITT population. The number of patients with response and responder rate, along with an exact two-sided 95% CI were summarized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 22
Percentage of Participants | 95.5 [77.2 to 99.9]
Statistical Analysis 1: Comparison: Eculizumab; Test type: Superiority or Other; Percent of Platelet Count Normalization = 95, 95% CI 2-sided [77.2 to 99.9]

4. Secondary Outcome: Proportion of Patients With Estimated Glomerular Filtration Rate (eGFR) Improvement
Description: Proportion of Patients with Estimated Glomerular Filtration Rate (eGFR) Improvement was determined and defined as an increase in eGFR by ≥ 15 mL/min/1.73m2 from baseline, sustained for at least two consecutive measurements obtained at least four weeks apart.
Time Frame: Through 26 weeks
Population: The tabulations of the proportions of patients with Estimated Glomerular Filtration Rate (eGFR) Improvement through 26 weeks were performed for the ITT population. The number of patients with response and responder rate, along with an exact two-sided 95% CI were summarized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 22
Percentage of Participants | 86.4 [65.1 to 97.1]
Statistical Analysis 1: Comparison: Eculizumab; Test type: Superiority or Other; Percent of eGFR Improvement = 86.4, 95% CI 2-sided [65.1 to 97.1]

5. Secondary Outcome: Platelet Count Change From Baseline to 26 Weeks
Time Frame: Through 26 weeks
Population: Change from baseline platelet counts were analyzed for the ITT population using a repeated measures ANOVA model. The estimated LS means of change from baseline at each post-baseline visit alongside with 95% CIs and P-values were calculated, as were the parameter estimates for the covariates and their associated P-values.
Measure: Least Squares Mean (95% Confidence Interval); unit: 10^9 cells/L
Arm/Group | Eculizumab
Number analyzed (Participants) | 22
10^9 cells/L | 204.96 [164.44 to 245.49]
Statistical Analysis 1: Comparison: Eculizumab; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean change from baseline = 204.96, 95% CI 2-sided [164.44 to 245.49]

6. Secondary Outcome: Proportion of Patients With Complete TMA Response
Description: as for outcome 1
Time Frame: Through End of Study, Median Exposure 55 Weeks
Population: The tabulations of the proportions of patients with Complete TMA Response through end of study were performed for the ITT population. Exact binomial two-sided 95% CI using the Clopper-Pearson method for the responder rate was presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 22
Percentage of Participants | 68.2 [45.1 to 86.1]
Statistical Analysis 1: Comparison: Eculizumab; Test type: Superiority or Other; Percent of Complete TMA Response = 68.2, 95% CI 2-sided [45.1 to 86.1]

7. Secondary Outcome: Proportion of Patients With Complete Hematologic Response
Description: Proportion of Patients with Complete Hematologic response through end of study was determined and defined by normalization of platelet count and LDH sustained for at least two consecutive measurements obtained at least four weeks apart.
Time Frame: Through End of Study, Median Exposure 55 Weeks
Population: The tabulations of the proportions of patients with Complete Hematologic Response through end of study were performed for the ITT population. The number of patients with response and responder rate, along with an exact two-sided 95% CI were summarized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 22
Percentage of Participants | 90.9 [70.8 to 98.9]
Statistical Analysis 1: Comparison: Eculizumab; Test type: Superiority or Other; Percent of Complete Hematologic Response = 90.9, 95% CI 2-sided [70.8 to 98.9]

8. Secondary Outcome: Proportion of Patients With Platelet Count Normalization
Description: Proportion of Patients with Platelet Count Normalization through end of study was determined and defined as the platelet count observed to be ≥ 150 x 109/L on at least two consecutive measurements which span a period of at least four weeks
Time Frame: Through End of Study, Median Exposure 55 Weeks
Population: The tabulations of the proportions of patients with Platelet Count Normalization through end of study were performed for the ITT population. The number of patients with response and responder rate, along with an exact two-sided 95% CI were summarized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 22
Percentage of Participants | 95.5 [77.2 to 99.9]
Statistical Analysis 1: Comparison: Eculizumab; Test type: Superiority or Other; Percent of Platelet Count Normalization = 95.5, 95% CI 2-sided [77.2 to 99.9]

9. Secondary Outcome: Proportion of Patients With Estimated Glomerular Filtration Rate (eGFR) Improvement
Description: as for outcome 4
Time Frame: Through End of Study, Median Exposure 55 Weeks
Population: The tabulations of the proportions of patients with eGFR Improvement through end of study were performed for the ITT population. The number of patients with response and responder rate, along with an exact two-sided 95% CI were summarized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 22
Percentage of Participants | 86.4 [65.1 to 97.1]
Statistical Analysis 1: Comparison: Eculizumab; Test type: Superiority or Other; Percent of eGFR Improvement = 86.4, 95% CI 2-sided [65.1 to 97.1]

10. Secondary Outcome: Platelet Count Change From Baseline to 52 Weeks
Time Frame: Through 52 Weeks
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: 10^9 cells/L
Arm/Group | Eculizumab
Number analyzed (Participants) | 22
10^9 cells/L | 165.43 [98.43 to 232.46]
Statistical Analysis 1: Comparison: Eculizumab; Test type: Superiority or Other; p < 0.0001, ANOVA; LS mean change from baseline = 165.43, 95% CI 2-sided [98.43 to 232.43]

11. Secondary Outcome: Pharmacokinetics (PK) and Pharmacodynamics (PD); Minimum and Maximum Blood Concentration (Body Weight Cohort 5 - <10kg) N=3
Time Frame: Induction Phase was between 1 and 4 weeks in length depending on patient weight cohort.Maintenance Phase was started 1 week after induction phase and dosing of eculizumab administration was every 2 weeks or every 3 weeks depending on patient weight cohort
Population: PK parameters Cmin and Cmax were estimated using a population PK model developed from the observed PK concentration data
Measure: Mean (Standard Deviation); unit: micrograms/mL
Groups:
- Eculizumab. Min and Max Blood Concentration: 5 - <10kg weight cohort
Arm/Group | Eculizumab. Min and Max Blood Concentration
Number analyzed (Participants) | 3
micrograms/mL
  Min Concentration during induction period | 223.2 (19.0)
  Max concentration during induction period | 312.8 (51.2)
  Min concentration during maintenance | 187.2 (42.0)
  Max concentration during maintenance | 499.7 (27.8)

12. Secondary Outcome: Pharmacokinetics (PK) and Pharmacodynamics (PD); Minimum and Maximum Blood Concentration (Body Weight Cohort 10 - <20kg) N=7
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms/mL
Groups:
- Eculizumab. Min and Max Blood Concentration: 10 - <20kg weight cohort
Arm/Group | Eculizumab. Min and Max Blood Concentration
Number analyzed (Participants) | 7
micrograms/mL
  Min Concentration during induction period | 297.2 (74.7)
  Max concentration during induction period | 436.3 (128.3)
  Min concentration during maintenance | 241.8 (106.0)
  Max concentration during maintenance | 459.5 (105.5)

13. Secondary Outcome: Pharmacokinetics (PK) and Pharmacodynamics (PD); Minimum and Maximum Blood Concentration (Body Weight Cohort 20 - <30kg)
Time Frame: Induction Phase was between 1 and 4 weeks in length depending on patient weight cohort. Maintenance Phase was started either 2 weeks or 3 weeks after induction phase depending on patient weight cohort
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms/mL
Groups:
- Eculizumab. Min and Max Blood Concentration: 20 - <30kg weight cohort
Arm/Group | Eculizumab. Min and Max Blood Concentration
Number analyzed (Participants) | 6
micrograms/mL
  Min Concentration during induction period | 185.1 (19.5)
  Max concentration during induction period | 242.5 (24.5)
  Min concentration during maintenance | 337.6 (43.4)
  Max concentration during maintenance | 579.5 (66.5)

14. Secondary Outcome: Pharmacokinetics (PK) and Pharmacodynamics (PD); Minimum and Maximum Blood Concentration (Body Weight Cohort 30 - <40kg) N=1
Time Frame: as for outcome 13
Population: PK parameters Cmin and Cmax were estimated using a population PK model developed from the observed PK concentration data. N=0 in the maintenance phase because the patient changed to ≥40kg body weight category
Measure: Mean (Standard Deviation); unit: micrograms/mL
Groups:
- Eculizumab. Min and Max Blood Concentration: 30 - <40kg weight cohort
Arm/Group | Eculizumab. Min and Max Blood Concentration
Number analyzed (Participants) | 1
micrograms/mL
  Min Concentration during induction period | 196.8
  Max concentration during induction period | 282.2
  Min concentration during Maintenance | NA (NA) — N=6 in the maintenance phase because the patient in the 30 - <40kg cohort group changed to the ≥40kg body weight category
  Max concentration during Maintenance | NA (NA) — N=6 in the maintenance phase because the patient in the 30 - <40kg cohort group changed to the ≥40kg body weight category

15. Secondary Outcome: Pharmacokinetics (PK) and Pharmacodynamics (PD); Minimum and Maximum Blood Concentration (Body Weight Cohort ≥40kg) N=5
Time Frame: as for outcome 13
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms/mL
Groups:
- Eculizumab. Min and Max Blood Concentration: ≥40kg weight cohort
Arm/Group | Eculizumab. Min and Max Blood Concentration
Number analyzed (Participants) | 5
micrograms/mL
  Min Concentration during induction period | 125.5 (26.3)
  Max concentration during induction period | 180.9 (42.6)
  Min concentration during maintenance | 278.4 (130.3)
  Max concentration during maintenance | 572.8 (267.7)

ADVERSE EVENTS:
Time Frame: Through end of study; exposure to eculizumab in this study extended for a median duration of 12.6 months and ranged from 1 dose to 24.5 months.
Description: At every visit, patients were asked a standard non-leading question to elicit any changes in their medical well-being including inquiry about any hospitalization, accidents and new or changed concomitant medication regimens. AEs were also documented from any data collected (e.g. laboratory values, physical examination findings, ECG changes, etc.)
Arm/Group | Eculizumab
Serious Adverse Events (participants affected / at risk) | 13/22
Other Adverse Events (participants affected / at risk) | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=22)
Anaemia (Blood and lymphatic system disorders) | 2
Bone marrow failure (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Device malfunction (General disorders) | 1
Medical device complication (General disorders) | 1
Pyrexia (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Device related sepsis (Infections and infestations) | 1
Enterocolitis viral (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 2
Infection (Infections and infestations) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 2
Overdose (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Metabolic disorder (Metabolism and nutrition disorders) | 1
Agitation (Psychiatric disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Uterine polyp (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=22)
ANAEMIA (Blood and lymphatic system disorders) | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 1
LYMPHOPENIA (Blood and lymphatic system disorders) | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 1
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 2
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 1
EAR PAIN (Ear and labyrinth disorders) | 1
HYPOTHYROIDISM (Endocrine disorders) | 1
EYE DISCHARGE (Eye disorders) | 1
ULCERATIVE KERATITIS (Eye disorders) | 1
VISION BLURRED (Eye disorders) | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 7
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2
CONSTIPATION (Gastrointestinal disorders) | 2
DIARRHOEA (Gastrointestinal disorders) | 8
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1
DYSPEPSIA (Gastrointestinal disorders) | 3
DYSPHAGIA (Gastrointestinal disorders) | 1
GASTRITIS (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 7
ASTHENIA (General disorders) | 1
APPLICATION SITE ECZEMA (General disorders) | 1
CHEST PAIN (General disorders) | 1
DRUG WITHDRAWAL SYNDROME (General disorders) | 1
FATIGUE (General disorders) | 1
INJECTION SITE RASH (General disorders) | 1
INJECTION SITE HAEMATOMA (General disorders) | 2
MALAISE (General disorders) | 1
PAIN (General disorders) | 1
OEDEMA PERIPHERAL (General disorders) | 1
PYREXIA (General disorders) | 11
ACUTE TONSILLITIS (Infections and infestations) | 2
BETA HAEMOLYTIC STREPTOCOCCAL INFECTION (Infections and infestations) | 1
BRONCHITIS (Infections and infestations) | 1
CANDIDURIA (Infections and infestations) | 1
CATHETER SITE INFECTION (Infections and infestations) | 3
CONJUNCTIVITIS VIRAL (Infections and infestations) | 1
EAR INFECTION (Infections and infestations) | 1
ESHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1
FUNGAL INFECTION (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 2
GENITAL CANDIDIASIS (Infections and infestations) | 1
INFLUENZA (Infections and infestations) | 1
NASOPHARYNGITIS (Infections and infestations) | 7
ORAL FUNGAL INFECTION (Infections and infestations) | 1
OTITIS MEDIA (Infections and infestations) | 1
PHARYNGITIS (Infections and infestations) | 1
PATHOGEN RESISTANCE (Infections and infestations) | 1
PYELONEPHRITIS (Infections and infestations) | 1
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1
RHINITIS (Infections and infestations) | 5
SINUSITIS (Infections and infestations) | 1
SKIN INFECTION (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7
URINARY TRACT INFECTION (Infections and infestations) | 4
VARICELLA (Infections and infestations) | 1
VIRAL INFECTION (Infections and infestations) | 2
ANIMAL BITE (Injury, poisoning and procedural complications) | 1
CONTUSION (Injury, poisoning and procedural complications) | 2
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1
SCRATCH (Injury, poisoning and procedural complications) | 2
BLOOD BICARBONATE DECREASED (Investigations) | 1
ELECTROCARDIOGRAM T WAVE INVERSION (Investigations) | 1
ELECTROENCEPHALOGRAM ABNORMAL (Investigations) | 1
WEIGHT INCREASED (Investigations) | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1
METABOLIC DISORDER (Metabolism and nutrition disorders) | 1
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 3
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
DEMYELINATING POLYNEUROPATHY (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 5
SINUS HEADACHE (Nervous system disorders) | 1
FOOD AVERSION (Psychiatric disorders) | 1
MOOD ALTERED (Psychiatric disorders) | 1
CALCULUS URINARY (Renal and urinary disorders) | 1
DYSURIA (Renal and urinary disorders) | 1
PROTEINURIA (Renal and urinary disorders) | 1
GLYCOSURIA (Renal and urinary disorders) | 1
MICROALBUMINURIA (Renal and urinary disorders) | 1
POLYURIA (Renal and urinary disorders) | 1
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 9
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1
TONSILLAR HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 3
DERMATITIS DIAPER (Skin and subcutaneous tissue disorders) | 2
ECZEMA (Skin and subcutaneous tissue disorders) | 1
INCREASED TENDENCY TO BRUISE (Skin and subcutaneous tissue disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1
PURPURA (Skin and subcutaneous tissue disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 4
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 1
SKIN LESION (Skin and subcutaneous tissue disorders) | 1
HAEMATOMA (Vascular disorders) | 2
HYPERTENSION (Vascular disorders) | 4
PALLOR (Vascular disorders) | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 1
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
NAIL INJURY (Injury, poisoning and procedural complications) | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1
CENTRAL VENOUS CATHETER REMOVAL (Surgical and medical procedures) | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Participation in this multicenter study involved a commitment to publish the data from the study in a cooperative publication prior to release of study results on an individual basis.